CLINICAL TRIAL: NCT05198193
Title: Evaluation and Development of Falls Prevention and Management in the Community of Central and North of Singapore for Older Adults
Brief Title: Evaluation and Development of Falls Prevention and Management in the Community for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Noah Lim, Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NUS-IRB-2020-024
Record Dates: First submitted 2021-12-07; First posted 2022-01-20 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Falls Risk; Falls Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control - Older Adults (Experimental): Participants age 60 years old or above.
  Interventions: Behavioral: No Message Given
- Positive - Older Adults (Experimental): Participants age 60 years old or above.
  Interventions: Behavioral: Positive Message Given - Older Adults
- Negative - Older Adults (Experimental): Participants age 60 years old or above.
  Interventions: Behavioral: Negative Message Given - Older Adults
- Control - Younger Adults (Experimental): Participants age between 30 and 59 years old.
  Interventions: Behavioral: No Message Given
- Positive - Younger Adults (Experimental): Participants age between 30 and 59 years old.
  Interventions: Behavioral: Positive Message Given - Younger Adults
- Negative - Younger Adults (Experimental): Participants age between 30 and 59 years old.
  Interventions: Behavioral: Negative Message Given - Younger Adults

INTERVENTIONS:
Behavioral: No Message Given — Participants in this arm are not given any intervention.
  Arms: Control - Older Adults; Control - Younger Adults
Behavioral: Positive Message Given - Older Adults — Participants in this arm are given a positively framed message from an older adult's point of view.
  Arms: Positive - Older Adults
Behavioral: Negative Message Given - Older Adults — Participants in this arm are given a negatively framed message from an older adult's point of view.
  Arms: Negative - Older Adults
Behavioral: Positive Message Given - Younger Adults — Participants in this arm are given a positively framed message from an adult child's point of view.
  Arms: Positive - Younger Adults
Behavioral: Negative Message Given - Younger Adults — Participants in this arm are given a negatively framed message from an adult child's point of view.
  Arms: Negative - Younger Adults

SUMMARY:
This study investigates how differently-framed messages can affect people's attitude towards falls risk and prevention in older adults. This study considers the potentiality of adult children acting as change agents in influencing parents in falls prevention.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) will be conducted to test the effectiveness of two messaging types (positively vs negatively framed) via two target audiences (older vs younger adults).

The RCT evaluates the effectiveness of the differently-framed messages delivered to older and younger adults in affecting people's attitude toward falls risk and motivating them to learn about preventing falls. Also, the potential of adult children acting as change agents to positively influence parents in preventing falls is explored.

Older and younger adults who are eligible to participate in this study are randomly given one message. For older adults, the objective is to study which message is more effective in affecting their attitude towards falls risk and motivating them to learn about preventing falls. For younger adults, the aim is to understand which message is more effective in motivating them to learn about preventing falls for their parents.

Hypotheses:

H1: The negatively framed message is more effective than the positively framed counterpart in motivating older adults to find out about preventing falls. However, this effect decreases as the socioeconomic status decreases.

H2: The negatively framed message is more effective than the positively framed counterpart in motivating younger adults to find out about preventing falls.

ELIGIBILITY:
Inclusion Criteria:

* Singaporean or Permanent Residents (PRs)
* Read/speak English, Mandarin, or Malay
* Either age 60 years old and above, walk independently with or without assistive devices, have no self-reported/detected dementia or cognitive impairments or age between 30 and 59 years old and have either one of the parents age 60 years old and above who walk independently with or without assistive devices

Exclusion Criteria:

* Not Singaporean or PRs
* Do not read/speak English, Chinese, and Malay
* Age 29 years old and below
* Cannot walk independently with and without assistive devices
* Have self-reported/detected dementia or cognitive impairments

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
How much does the participant want to find out about preventing falls for himself/herself or his/her father/mother? | After being given a message during the survey, an average of 2 minutes
  This is a scale variable ranging from 1 to 9, which is "1" if not at all and "9" if a lot

SECONDARY OUTCOMES:
Whether the participant or the participant's father/mother has fallen in the past 12 months | After being given a message during the survey, an average of 2 minutes
  This is a categorical variable, which is "Yes" if the participant or the participant's father/mother has fallen in the past 12 months, "No" if not, and "Do not know" if the participant does not know whether his/her father/mother has fallen in the past 12 months
Whether the participant or the participant's father/mother is concerned about falling | After being given a message during the survey, an average of 2 minutes
  This is a categorical variable, which is "Very concerned" if the participant or the participant's father/mother is very concerned about falling, "Slightly concerned" if s/he is slightly concerned about falling, "Not concerned" if s/he is not concerned about falling, and "Do not know" if the participant does not know whether his/her father/mother is concerned about falling
Whether the participant or the participant's father/mother feels like s/he is going to fall when standing or walking | After being given a message during the survey, an average of 2 minutes
  This is a categorical variable, which is "Always" if the participant or the participant's father/mother always feels like s/he is going to fall when standing or walking, "Sometimes" if s/he sometimes feels like s/he is going to fall when standing or walking, "Never" if s/he never feels like s/he is going to fall when standing or walking, and "Do not know" if the participant does not know whether his/her father/mother feels like s/he is going to fall when standing or walking

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lim, PhD, Study Director — The Global Asia Institute, The National University of Singapore; Tuo-Yu Chen, PhD, Principal Investigator — Master Program in Global Health and Development, Taipei Medical University; Su-Chin Hsu, PhD, Principal Investigator — The Global Asia Institute, The National University of Singapore; Lianjun Li, PhD, Principal Investigator — The Global Asia Institute, The National University of Singapore; Catherine Yeung, PhD, Principal Investigator — Department of Marketing, The Chinese University of Hong Kong
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickinson A, Machen I, Horton K, Jain D, Maddex T, Cove J. Fall prevention in the community: what older people say they need. Br J Community Nurs. 2011 Apr;16(4):174-80. doi: 10.12968/bjcn.2011.16.4.174. PMID 21471918
- [Background] Liu X, Shuster MM, Mikels JA, Stine-Morrow EAL. Doing What Makes You Happy: Health Message Framing for Younger and Older Adults. Exp Aging Res. 2019 Jul-Sep;45(4):293-305. doi: 10.1080/0361073X.2019.1627491. Epub 2019 Jun 12. PMID 31188722